CLINICAL TRIAL: NCT04980378
Title: Post Approval Study Protocol for the Two Level Simplify® Cervical Artificial Disc
Status: Completed | Type: Observational
Sponsor: NuVasive (Industry)
Responsible Party: Sponsor
Organization: Globus Medical Inc (Industry)
Other Study IDs: P200022_S003_PAS
Record Dates: First submitted 2021-07-19; First posted 2021-07-28 (Actual); Results first posted 2025-03-26 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Cervical Degenerative Disc Disorder
Keywords: Two Level

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Simplify Disc: Extended follow-up of IDE Subjects treated at two continuous levels with the Simplify Cervical Artificial Disc during IDE G150206
  Interventions: Device: Simplify Disc
- Historical Control - Anterior Cervical Discectomy and Fusion (ACDF): This study used a non-concurrent historical control with subject-level data on a parallel group design. The historical control group was formed from the randomized ACDF arm of a previously completed two level cervical disc trial.

INTERVENTIONS:
Device: Simplify Disc — The Simplify Disc is a cervical artificial disc manufactured from polyether ether ketone (PEEK) endplates and a mobile, zirconia-toughened alumina ceramic core.
  Groups: Simplify Disc

SUMMARY:
This study is intended to demonstrate the 5-year long-term safety and efficacy of the Simplify® Cervical Artificial Disc ("Simplify Disc") in subjects enrolled in the non-randomized two-level Simplify Disc Investigational Device Exemption (IDE) study. This study was conducted under IDE G150206

ELIGIBILITY:
Inclusion Criteria:

- All subjects enrolled in the two level Simplify Disc IDE study are considered for this long-term follow-up study.

Exclusion Criteria:

* Subjects who were not implanted with the Simplify Disc during the IDE study
* Subjects who had a secondary surgical intervention at the index level during the IDE study
* Subjects who were withdrawn or withdrew consent to participate in the IDE study
* Subjects who do not consent to participate in long-term follow-up post-approval study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will include subjects who were enrolled in the IDE study G150206. This will include up to 170 subjects eligible for study enrollment from sixteen (16) sites in the two level Simplify Disc IDE study who consent to long-term follow-up. Additionally, up to 17 training subjects from the two level Simplify Disc IDE study from seventeen (17) sites will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 291 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2024-01-24 (Actual); Study Completion 2024-01-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kyle Malone, Study Director — Globus Medical
Locations (18):
- United States (18):
  - Orthopaedic Education and Research Institute of Southern California, Orange, California
  - The Spine Institute for Spine Restoration, Santa Monica, California
  - Spine Education and Research Foundation, Thornton, Colorado
  - Connecticut Orthopaedic Specialists, Hamden, Connecticut
  - Kennedy-White Orthopedic Center, Sarasota, Florida
  - NorthShore University Health System, Evanston, Illinois
  - Indiana Spine Group, Carmel, Indiana
  - Parkview Research Center, Fort Wayne, Indiana
  - Orthopaedic Institute of Western Kentucky, Paducah, Kentucky
  - Spine Institute of Louisiana, Shreveport, Louisiana
  - William Beaumont Hospital Research Institute, Royal Oak, Michigan
  - Buffalo Spine Surgery, Lockport, New York
  - Carolina Neurosurgery and Spine Associates, Charlotte, North Carolina
  - Oregon Neurosurgery, Springfield, Oregon
  - Texas Spine Consultants, Addison, Texas
  - Texas Back Institute, Plano, Texas
  - The Disc Replacement Center, West Jordan, Utah
  - Virginia Spine Institute, Reston, Virginia

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: No recruitment - long term follow up of subjects previously enrolled in Investigational Device Exemption (IDE) and historical control data
Groups:
- Historical ACDF Control: A non-concurrent historical control was used with subject-level data on a parallel group design. The historical control group was formed from the randomized ACDF arm of a previously completed two-level cervical disc IDE trial. (Note: sponsor is unable to disclose NCT number of historical study due to contractual obligations)
Period: Overall Study
Arm/Group | Simplify Disc | Historical ACDF Control
Started | 157 | 134 (Historical data)
Completed | 144 | 107 (Historical data)
Not Completed | 13 | 27

BASELINE CHARACTERISTICS:
Groups:
- Historical ACDF Control: Historical ACDF Data from similar protocol used as control.
- Total: Total of all reporting groups
Arm/Group | Simplify Disc | Historical ACDF Control | Total
Number analyzed (Participants) | 157 | 134 | 291
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.35 (9.04) | 47.71 (7.83) | 48.59 (8.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83 | 71 | 154
  Male | 74 | 63 | 137
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 6 | 11
  White | 146 | 122 | 268
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 3 | 8
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 157 | 134 | 291

OUTCOME MEASURES:

1. Primary Outcome: Clinical Composite Success
Description: Individual success for Simplify Disc was defined as follows:
  * Neck Disability Index (NDI) score improvement of at least 15 points from pre-operative;
  * Maintenance or improvement in neurological status;
  * No serious adverse event classified as implant associated or implant/surgical procedure associated; and
  * No additional surgical procedure classified as a "failure."
Time Frame: Data through 24 months gathered in IDE (NCT03123549; start date 4/1/17). This PAS (start date 8/1/21) followed the same patient cohort through 60 months post-op. Comparison data from historical controls up to 60 months post-op is also reported
Population: While 144 Simplify Disc subjects completed the 60-month visit, 140 Simplify Disc subjects had completed change in Neck Disability Index and neurologic data at 60 months due to missed questionnaires and/or neurologic exams.
Measure: Count of Participants; unit: Participants
Groups:
- ACDF: Historical ACDF control data: Historical ACDF Data from similar protocol used as control.
Arm/Group | Simplify Disc | ACDF: Historical ACDF control data
Number analyzed (Participants) | 140 | 107
Participants | 127 | 84

2. Secondary Outcome: Clinically Significant Improvement in One or More Radicular Symptoms or Myelopathy
Description: An arm pain questionnaire was used to measure radicular symptoms and compare to baseline symptoms in the IDE study. Changes of at least 2 points on a 10-point scale were regarded as clinically significant (0=no pain; 10=worst pain)
Time Frame: as for outcome 1
Population: While 144 Simplify Disc subjects completed the 60-month visit, 136 subjects had change in Arm Pain Intensity data at 60 months due to missed questionnaires. Likewise, 107 ACDF control subjects completed the 60-month visit, but 104 had change in Arm Pain Intensity data at 60 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Simplify Disc | ACDF: Historical ACDF control data
Number analyzed (Participants) | 136 | 104
Participants | 125 | 90

3. Secondary Outcome: Health Survey; 36-Item Short Form Survey (SF-36) - Physical Component Score (PCS) Maintenance or Improvement
Description: The PCS is a sub-score of the SF-36. The SF-36 is a multipurpose survey with 36 questions. The questions were combined, scored, and weighted to create two scores that provide glimpses into mental and physical functioning and overall health-related quality-of-life. Higher scores indicate better outcomes. Scores range from 0-50. Maintenance or improvement was defined as PCS(Postop) - PCS(Preop) ≥0.
Time Frame: as for outcome 1
Population: While 144 Simplify Disc subjects completed the 60-month visit, 135 Simplify Disc subjects had SF-36 data available at 60 months due to missed questionnaires. Likewise, 107 ACDF subjects completed the 60-month visit, but 104 had SF-36 data available at 60 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Simplify Disc | ACDF: Historical ACDF control data
Number analyzed (Participants) | 135 | 104
Participants
  Maintenance or improvement | 122 | 86
  Absence of maintenance or improvement | 13 | 18

4. Secondary Outcome: Health Survey; 36-Item Short Form Survey (SF-36) - Mental Component Score (MCS) Maintenance or Improvement
Description: The MCS is a sub-score of the SF-36. The SF-36 is a multipurpose survey with 36 questions. The questions were combined, scored, and weighted to create two scores that provide glimpses into mental and physical functioning and overall health-related quality-of-life. Higher scores indicate better outcomes. Scores range from 0-50. Maintenance or improvement was defined as PCS(Postop) - PCS(Preop) ≥0.
Time Frame: as for outcome 1
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Simplify Disc | ACDF: Historical ACDF control data
Number analyzed (Participants) | 135 | 104
Participants
  Maintenance or improvement | 110 | 80
  Absence of maintenance or improvement | 25 | 24

5. Secondary Outcome: Dysphagia Handicap Index (DHI Scale)
Description: Dysphagia Handicap Index score for the Simplify Disc subjects at 60 months. A higher score is indicative of a less desirable outcome. It is scored 0-100.
  Data was not collected on DHI in the historical ACDF control group. Only Simplify Disc subjects are reported. This was pre-specified in the study design.
Time Frame: Data through 24 months gathered in IDE (NCT03123549 with start date of 4/1/17). This PAS (start date 8/1/21) followed the same patient cohort through 60 months post-operative.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Simplify Disc
Number analyzed (Participants) | 144
score on a scale | 7.1 (11.6)

6. Secondary Outcome: Patient Satisfaction
Description: Patient satisfaction was assessed by survey based on the response to the statement "I am satisfied with the results of my surgery" at 60 months. Answer options ranged from definitely true to definitely false.
Time Frame: as for outcome 1
Population: While 144 Simplify Disc subjects completed the 60-month visit, 143 subjects had evaluable treatment satisfaction data at 60 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Simplify Disc | ACDF: Historical ACDF control data
Number analyzed (Participants) | 143 | 107
Participants
  Definitely true | 116 | 77
  Mostly true | 22 | 24
  Don't know | 3 | 4
  Mostly false | 2 | 1
  Definitely false | 0 | 1

7. Secondary Outcome: Physician's Perception
Description: Results at 60 months were categorized by the physician's perception of the subject's condition (excellent, good, fair, or poor).
Time Frame: as for outcome 1
Population: While 144 Simplify Disc subjects completed the 60-month visit, 141 subjects had evaluable Physician's Perception of Results data at 60 months due to missed questionnaires.
Measure: Count of Participants; unit: Participants
Arm/Group | Simplify Disc | ACDF: Historical ACDF control data
Number analyzed (Participants) | 141 | 107
Participants
  Excellent | 126 | 57
  Good | 10 | 41
  Fair | 5 | 8
  Poor | 0 | 1

8. Secondary Outcome: Change in Average Disc Height (Superior Index Level)
Description: Average disc height (superior index level) at 60 months was compared to the baseline measurement in the IDE study and the change was calculated. Measurements were scored by an independent core lab. Average disc height was calculated as the simple average of the anterior and posterior disc heights.
  Data was not collected on average disc height in the historical ACDF control group. Only Simplify Disc subjects are reported. This was pre-specified in the study design.
Time Frame: as for outcome 5
Population: While 144 Simplify Disc subjects completed the 60-month visit, 140 subjects had evaluable radiographs for this assessment at 60 months due to missed x-rays or poor image quality which limited analysis.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Simplify Disc
Number analyzed (Participants) | 140
mm | 1.10 (0.84)

9. Secondary Outcome: Change in Average Disc Height (Inferior Index Level)
Description: Average disc height (inferior index level) at 60 months was compared to the baseline measurement in the IDE study and the change was calculated. Measurements were scored by an independent core lab. Average disc height was calculated as the simple average of the anterior and posterior disc heights.
  Data was not collected on average disc height in the historical ACDF control group. Only Simplify Disc subjects are reported. This was pre-specified in the study design.
Time Frame: as for outcome 5
Population: While 144 Simplify Disc subjects completed the 60-month visit, 131 subjects had evaluable radiographs for this assessment at 60 months due to missed x-rays or poor image quality which limited analysis.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Simplify Disc
Number analyzed (Participants) | 131
mm | 0.81 (0.94)

10. Secondary Outcome: Adjacent Level Deterioration - Superior Adjacent Level
Description: Outcome reports the number and percentage of subjects with adjacent level disc degeneration (ALDD) above the index level based on X-ray images. Degeneration was graded as none (no degenerative changes), doubtful (Minimal osteophytosis only), minimal (Definite osteophytosis with some sclerosis of anterior part of vertebral plates), moderate (Marked osteophytosis and sclerosis of vertebral plates with slight narrowing of disk space), or severe (Large osteophytes, marked sclerosis of vertebral plates, and marked narrowing of disk space). Assessments were made by an independent core lab.
  Data was not collected on adjacent level deterioration in the historical ACDF control group. Only Simplify Disc subjects are reported. This was pre-specified in the study design.
Time Frame: as for outcome 5
Population: While 144 Simplify Disc subjects completed the 60-month visit, 137 Simplify Disc subjects had evaluable radiographs for this assessment at 60 months due to missed x-rays or poor image quality which limited analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Simplify Disc
Number analyzed (Participants) | 137
Participants
  None | 70
  Doubtful | 41
  Minimal | 20
  Moderate | 5
  Severe | 1

11. Secondary Outcome: Adjacent Level Deterioration - Inferior Adjacent Level
Description: Outcome reports the number and percentage of subjects with adjacent level disc degeneration (ALDD) below the index level based on X-ray images. Degeneration was graded as none (no degenerative changes), doubtful (Minimal osteophytosis only), minimal (Definite osteophytosis with some sclerosis of anterior part of vertebral plates), moderate (Marked osteophytosis and sclerosis of vertebral plates with slight narrowing of disk space), or severe (Large osteophytes, marked sclerosis of vertebral plates, and marked narrowing of disk space). Assessments were made by an independent core lab.
  Data was not collected on adjacent level deterioration in the historical ACDF control group. Only Simplify Disc subjects are reported. This was pre-specified in the study design.
Time Frame: as for outcome 5
Population: While 144 Simplify Disc subjects completed the 60-month visit, 124 Simplify Disc subjects had evaluable radiographs for this assessment at 60 months due to missed x-rays or poor image quality which limited analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Simplify Disc
Number analyzed (Participants) | 124
Participants
  None | 81
  Doubtful | 23
  Minimal | 13
  Moderate | 5
  Severe | 2

12. Secondary Outcome: Displacement or Migration of the Device
Description: Displacement or migration of the device at 60 months was be compared to immediate post-op data collected in the IDE study. This was be graded by the radiographic core lab. Migration was considered "present" if changes of >3mm were noted. The superior index level and inferior index level was assessed separately.
Time Frame: as for outcome 1
Population: While 144 Simplify Disc subjects completed the 60-month visit, 140 subjects had evaluable radiographs for this assessment at 60 months due to missed x-rays or poor image quality which limited analysis. Likewise, 107 ACDF subjects completed the 60-month visit, but 102 had 60-month radiographs available for this assessments.
Measure: Count of Participants; unit: Participants
Arm/Group | Simplify Disc | ACDF: Historical ACDF control data
Number analyzed (Participants) | 140 | 102
Participants
  Migration present at either index level | 0 | 0
  Migration absent at both index levels | 140 | 102

ADVERSE EVENTS:
Time Frame: Data presented includes adverse events (AEs) collected under both the parent IDE study (G150206) and this Post Approval Study (PAS) for patients who enrolled in this PAS. Data collected from the time of surgery through 24 months was gathered in the IDE (NCT03123549; start date 4/1/17) and data for the same patient cohort from 24 months through 60 months post-op was gather under this PAS (start date 8/1/21). Comparison data from historical controls through 60 months post-op is also reported
Description: All adverse events were reviewed and adjudicated by an independent Clinical Events Committee.
Arm/Group | Simplify Disc | ACDF: Historical ACDF Control Data
All-Cause Mortality (participants affected / at risk) | 0/157 | 0/134
Serious Adverse Events (participants affected / at risk) | 40/157 | 54/134
Other Adverse Events (participants affected / at risk) | 119/157 | 126/134
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Simplify Disc (N=157) | ACDF: Historical ACDF Control Data (N=134)
Lumbar radiculopathy (Musculoskeletal and connective tissue disorders) | 13 (14) | 14 (14)
Infection (not at surgical site) (Infections and infestations) | 7 (8) | 2 (2)
Appendicular arthritis (Musculoskeletal and connective tissue disorders) | 3 (4) | 6 (6)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 3 (3)
Other (General disorders) | 2 (2) | 4 (4)
Low back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (5)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 3 (3)
Accidental trauma (General disorders) | 3 (3) | 2 (2)
Gastrointestinal complications (Gastrointestinal disorders) | 2 (2) | 2 (2)
Cervical radiculopathy (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Pain (no narcotic given) (General disorders) | 2 (2) | 1 (1)
Hematoma or seroma (Vascular disorders) | 2 (2) | 0 (0)
Stroke (Vascular disorders) | 2 (2) | 0 (0)
Difficulty with urination (Renal and urinary disorders) | 1 (1) | 1 (1)
Embolism (Vascular disorders) | 1 (1) | 1 (1)
Inflammation (General disorders) | 1 (2) | 1 (1)
Blood loss (greater than 500 mL) (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Vertebral fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Thromboembolism (Vascular disorders) | 1 (1) | 0 (0)
Nonunion/pseudoarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (5)
Psychological illness (Psychiatric disorders) | 0 (0) | 3 (3)
Development of DDD at adjacent levels (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Surgery at a location other than the spine (Surgical and medical procedures) | 0 (0) | 2 (2)
Cerebrospinal fluid leakage (Nervous system disorders) | 0 (0) | 1 (1)
Coordination abnormalities (General disorders) | 0 (0) | 1 (1)
Headache (General disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pulmonary embolism (Vascular disorders) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Surgery at another spine level (Surgical and medical procedures) | 0 (0) | 1 (1)
Cardiac event (Cardiac disorders) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Soft tissue damage (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dermatitis/Skin allergy (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Low back pain (narcotic given) (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Renal dysfunction (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Simplify Disc (N=157) | ACDF: Historical ACDF Control Data (N=134)
Pain (no narcotic given) (General disorders) | 32 (38) | 37 (43)
Accidental trauma (General disorders) | 27 (30) | 39 (46)
Inflammation (General disorders) | 30 (39) | 29 (33)
Cervical radiculopathy (Musculoskeletal and connective tissue disorders) | 29 (38) | 29 (30)
Lumbar radiculopathy (Musculoskeletal and connective tissue disorders) | 30 (37) | 28 (28)
Appendicular arthritis (Musculoskeletal and connective tissue disorders) | 11 (12) | 32 (43)
Infection (not at surgical site) (Infections and infestations) | 22 (27) | 18 (22)
Compressive neuropathy (Nervous system disorders) | 18 (22) | 20 (20)
Headache (General disorders) | 8 (8) | 23 (23)
Other (General disorders) | 11 (13) | 19 (22)
Low back pain (no narcotic given) (Musculoskeletal and connective tissue disorders) | 10 (10) | 12 (12)
Pain (narcotic given) (General disorders) | 8 (10) | 11 (11)
Gastrointestinal complications (Gastrointestinal disorders) | 6 (6) | 21 (25)
Development of DDD at adjacent levels (Musculoskeletal and connective tissue disorders) | 1 (1) | 13 (13)
Low back pain (narcotic given) (Musculoskeletal and connective tissue disorders) | 1 (1) | 13 (13)
Non-Infectious pulmonary disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 12 (13)
Numbness - increased from pre-op or prior visit (Nervous system disorders) | 5 (5) | 11 (12)
Spasm (Musculoskeletal and connective tissue disorders) | 2 (2) | 11 (14)
Dysphagia (Gastrointestinal disorders) | 7 (7) | 9 (9)
Cardiac event (Cardiac disorders) | 4 (4) | 9 (11)
Neck stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 9 (9)
Psychological illness (Psychiatric disorders) | 3 (3) | 8 (12)
Hypertension (Vascular disorders) | 2 (2) | 8 (8)
Dermatitis/Skin allergy (Skin and subcutaneous tissue disorders) | 2 (2) | 8 (8)
Nonunion/pseudoarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 7 (7)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 7 (7)
Allergic rhinitis (Immune system disorders) | 0 (0) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication results vary per investigator and per clinical trial agreement.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-14): https://cdn.clinicaltrials.gov/large-docs/78/NCT04980378/Prot_SAP_000.pdf